CLINICAL TRIAL: NCT00802828
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Famotidine 40 mg Tablets Administered as 1 x 40 mg Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study Between Two Oral Formulations of Famotidine Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perrigo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40103
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Bioavailability
Keywords: bioavailability; famotidine
MeSH Terms: interventions — Famotidine

ARMS (2):
- Test Product (Active Comparator)
  Interventions: Drug: Famotidine Tablets, 40 mg
- Reference Product (Active Comparator)
  Interventions: Drug: Famotidine Tablets, 40 mg

INTERVENTIONS:
Drug: Famotidine Tablets, 40 mg

SUMMARY:
Compare the rate and extent of absorption of famotidine 40 mg tablets, administered as 1 x 40 mg tablet under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women 18 years of age or older
* body mass index below 30.0 kg/m2
* willing to participate and sin a copy of the informed consent form

Exclusion Criteria:

* recent history of drug or alcohol addiction or abuse
* pregnant or lactating women
* history of allergic response to heparin, famotidine, other H2-receptor antagonists, or other related drugs
* evidence of a clinically significant disorder or whose laboratory results were deemed to be clinically significant
* recipient of any drugs as part of a research study within 30 days prior to study dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed based on the pharmacokinetic variables, Cmax, AUCO-t and AUCO-infinity